CLINICAL TRIAL: NCT02268357
Title: Effects of Propranolol on Fear of Dental Extraction: Study Protocol for a Randomized Placebo-controlled Trial.
Brief Title: The Effects of Propranolol on Fear of Tooth or Molar Extraction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. J. de Lange, prof. dr. J. de Lange (mandated sponsor/principal investigator), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL42210.018.13
Record Dates: First submitted 2014-10-07; First posted 2014-10-20 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Dental Anxiety
Keywords: Dental Anxiety; Tooth Extraction; Propranolol
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): capsules PROPRANOLOL (study medication); 80 mg 1 hour preoperative; 40 mg directly postoperative
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): capsules MICROCRYSTALLINE CELLULOSE (study medication); 80 mg 1 hour preoperative; 40 mg directly postoperative
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Oral propranolol capsules
  Other Names: propranolol hydrochloride; propranolol HCl

SUMMARY:
Randomized, placebo-controlled, double-blind, parallel group clinical trial evaluating the anxiolytic effects of propranolol on fear of wisdom tooth removal. It is hypothesized that, compared to placebo, perioperative oral propranolol reduces dental trait anxiety at 1 month follow-up after wisdom tooth removal.

DETAILED DESCRIPTION:
RATIONALE Tooth and molar removals are among the most feared interventions in dentistry and oral and maxillofacial surgery (OMFS). Anxiety for these procedures not only produces discomfort to the patient, but may also induce patient behavior that impedes surgery, thereby increasing operative time and complicating postoperative recovery. In addition, it has been found that having undergone an extraction poses a significantly increased risk for developing chronic apprehension for dental surgical procedures, disproportionate forms of dental anxiety (i.e., dental phobia), and symptoms of post-traumatic stress. Addressing these problems effectively requires an intervention that reduces both state anxiety during surgery and dental trait anxiety in the long term.

OBJECTIVE The purpose of this trial is to determine the anxiolytic effects of the ß-adrenoreceptor antagonist propranolol on patients with high levels of fear in anticipation of dental extraction.

METHODS Trial design: Randomized, placebo-controlled, two-group, parallel, double-blind, single center trial of 34 participants. Population and recruitment: Consecutive patients, referred by their dentist to the department of Oral and Maxillofacial Surgery of the Academic Medical Center of the University Amsterdam, for at least two tooth and/or molar removals, with self-reported high to extreme fear in anticipation of dental extraction. Intervention: Two 40 mg propranolol capsules one hour prior to dental extraction, followed by one 40 mg capsule directly postoperatively. Comparator: Placebo capsules. Primary outcome: Dental trait anxiety score reduction from baseline to 4-weeks follow-up. Secondary outcomes: Self-reported anxiety during surgery; physiological parameters (heart rate and blood pressure) during recall of the crucial fear-related memory; self-reported vividness and emotional charge of the crucial fear-related memory.

RISKS AND BENEFITS ASSOCIATED WITH PARTICIPATION Participants of the trial will undergo regular dental extraction procedures (treatment as usual), with an additional potentially anxiolytic pharmacological intervention (propranolol) or placebo. The most important known side-effects of propranolol are mild and self-limiting.

ELIGIBILITY:
Inclusion criteria

1. Signed written informed consent
2. ≥ 18 Years of age on entry to the study
3. Self-reported high to extreme fear of tooth or molar removal
4. Dutch or English-speaking

Exclusion criteria

1. Asthma or other obstructive pulmonary disease
2. Cardiac failure
3. Cardiac arrhythmia
4. Renal failure
5. Insulin-dependent diabetes mellitus
6. Pregnant or breast-feeding
7. Current use of another ß-adrenoreceptor antagonist
8. Current use of anxiolytic or antidepressant medication
9. Currently in psychotherapy for dental anxiety
10. Systolic blood pressure < 100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 1 month follow-up in Short version of the Dental Anxiety Inventory (S-DAI) | Change from baseline at 1 month follow-up
  dental trait anxiety

SECONDARY OUTCOMES:
Change from baseline at 1 month follow-up in Self-reported vividness and emotional charge of the crucial fear-related memory | Change from Baseline at 1 month follow-up
  Visual analogue scale
Change from baseline at 1 month follow-up in State anxiety during treatment | Change from Baseline at 1 month follow-up
  Visual analogue scale
Change from baseline at 1 month follow-up in Physiological parameters (heart rate and blood pressure) during recall of the crucial fear-related memory | Change from Baseline at 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: prof. dr. J. de Lange, MD, DDS, PhD, Principal Investigator — Academic Medical Center (AMC) of Amsterdam; prof. dr. A. de Jongh, DDS, PhD, Study Director — Academic Center for Dentistry Amsterdam (ACTA), University of Amsterdam
Locations (1):
- Dept. of Oral and Maxillofacial Surgery, Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu HH, Milgrom P, Fiset L. Effect of a beta-adrenergic blocking agent on dental anxiety. J Dent Res. 1991 Sep;70(9):1306-8. doi: 10.1177/00220345910700091401. PMID 1918581
- [Background] Brunet A, Orr SP, Tremblay J, Robertson K, Nader K, Pitman RK. Effect of post-retrieval propranolol on psychophysiologic responding during subsequent script-driven traumatic imagery in post-traumatic stress disorder. J Psychiatr Res. 2008 May;42(6):503-6. doi: 10.1016/j.jpsychires.2007.05.006. Epub 2007 Jun 22. PMID 17588604
- [Background] Lonergan MH, Olivera-Figueroa LA, Pitman RK, Brunet A. Propranolol's effects on the consolidation and reconsolidation of long-term emotional memory in healthy participants: a meta-analysis. J Psychiatry Neurosci. 2013 Jul;38(4):222-31. doi: 10.1503/jpn.120111. PMID 23182304
- [Derived] Steenen SA, van Wijk AJ, van Westrhenen R, de Lange J, de Jongh A. Effects of propranolol on fear of dental extraction: study protocol for a randomized controlled trial. Trials. 2015 Nov 25;16:536. doi: 10.1186/s13063-015-1065-7. PMID 26607848